CLINICAL TRIAL: NCT00524277
Title: Phase II Trial of the HER2/Neu Peptide GP2 + GM-CSF Vaccine vs GM-CSF Alone in HLA-A2+ OR the Modified HER2/Neu Peptide AE37 + GM-CSF Vaccine vs GM-CSF Alone in HLA-A2- Node-Positive and High-Risk Node-Negative Breast Cancer Patients
Brief Title: Vaccine Therapy in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Collaborators: NuGenerex Immuno-Oncology (Industry); Norwell, Inc. (Industry)
Responsible Party: Principal Investigator, COL George Peoples, MD, FACS, Chief, Surgical Oncology, Brooke Army Medical Center; Director and Principal Investigator, Cancer Vaccine Development Program, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDR0000562261; BAMC-C.2007.098 (Other: BAMC Institutional Review Board); WRNMMC-20225 (Other: WRNMMC Institutional Review Board)
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): HLA-A2-positive patients receive GP2 peptide + GM-CSF vaccine intradermally (ID) every 3-4 weeks for a total of up to 6 inoculations.
  Interventions: Biological: GP2 peptide + GM-CSF vaccine
- Arm II (Active Comparator): HLA-A2-positive patients receive GM-CSF ID every 3-4 weeks for a total of up to 6 inoculations.
  Interventions: Biological: GM-CSF (sargramostim)
- Arm III (Experimental): HLA-A2-negative patients receive AE37 peptide/GM-CSF vaccine ID every 3-4 weeks for a total of up to 6 inoculations.
  Interventions: Biological: AE37 + GM-CSF vaccine
- Arm IV (Active Comparator): HLA-A2-negative patients receive GM-CSF ID ID every 3-4 weeks for a total of up to 6 inoculations
  Interventions: Biological: GM-CSF (sargramostim)

INTERVENTIONS:
Biological: GP2 peptide + GM-CSF vaccine — Given intradermally every 3-4 weeks for a total of up to 6 inoculations
  Other Names: GM-CSF (sargramostim)
  Arms: Arm I
Biological: GM-CSF (sargramostim) — GM-CSF given intradermally very 3-4 weeks for a total of up to 6 inoculations
  Arms: Arm II
Biological: AE37 + GM-CSF vaccine — Given intradermally every 3-4 weeks for a total of up to 6 inoculations
  Other Names: GM-CSF (sargramostim)
  Arms: Arm III
Biological: GM-CSF (sargramostim) — Given intradermally every 3-4 weeks for a total of up to 6 inoculations
  Arms: Arm IV

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells that express HER2/neu. Biological therapies, such as GM-CSF, may stimulate the immune system in different ways and stop tumor cells from growing. It is not yet known whether vaccine therapy is more effective than GM-CSF in treating breast cancer.

PURPOSE: This randomized phase II trial is studying vaccine therapy to see how well it works compared with GM-CSF in treating patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if the GP2 peptide/GM-CSF vaccine reduces the recurrence rate in HLA-A2-positive, HER2/neu-positive, node-positive, or high-risk node-negative breast cancer patients randomized to receive the vaccine versus the immunoadjuvant, sargramostim (GM-CSF), alone.
* To determine if the AE37 peptide/GM-CSF vaccine reduces the recurrence rate in HLA-A2-negative, HER2/neu-positive, node-positive or high-risk node-negative breast cancer patients randomized to receive the vaccine versus the immunoadjuvant, GM-CSF, alone.
* To monitor the invitro and invivo immunologic responses to the vaccines and correlate these responses with the clinical outcomes.
* To monitor for any unexpected toxicities with the vaccines.

OUTLINE: This is a multicenter study. Patients are stratified according to nodal status. Patients are randomized to 1 of 4 treatment arms.

* Arm I: HLA-A2-positive patients receive GP2 peptide/GM-CSF vaccine intradermally (ID) every 3-4 weeks for a total of up to 6 inoculations.
* Arm II: HLA-A2-positive patients receive solely GM-CSF ID
* Arm III: HLA-A2-negative patients receive AE37 peptide/GM-CSF vaccine ID every 3-4 weeks for a total of up to 6 inoculations.
* Arm IV: HLA-A2-negative patients receive solely GM-CSF ID

After completion of study therapy, patients are followed every 3 months for the first 24 months and then every 6 months for an additional 36 months.

Booster inoculations are administered at 12, 18, 24, and 30 months from the date of patients' enrollment into the study. One booster inoculation is administered at each timepoint (+/- 2 weeks) and will be the same inoculation (vaccine or GM-CSF only) as what patients received during their regular inoculation series.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

1. Lymph node-positive breast cancer or high-risk lymph node-negative breast cancer. The latter is defined by any one of the following criteria:

   * T2 disease
   * Grade 3 disease
   * Lymphovascular invasion
   * Estrogen receptor- or progesterone receptor-negative disease
   * HER2/neu-expressing tumor (immunohistochemistry [IHC] 3+ and/or amplified fluorescence in situ hybridization [FISH] >2.2, or N0 (i+))
2. HER2/neu-expressing tumor (IHC 1-3+ and or positive FISH >1.2)
3. Completion of primary standard of care breast cancer therapies (i.e., surgery, chemotherapy, immunotherapy and radiation therapy as appropriate per standard of care for patients' specific cancer)
4. Clinically cancer-free (no evidence of disease)
5. Patients may be enrolled between 1-6 months from completion of standard primary breast cancer therapies
6. Good performance status (as defined in Exclusion Criteria)
7. Capable of informed consent

Exclusion criteria:

1. HER2/neu-negative breast cancers (IHC 0)
2. Clinical and/or radiographic evidence of residual or persistent breast cancer
3. Receiving immunosuppressive therapy to include chemotherapy, steroids, or methotrexate
4. In poor health (Karnofsky <60%, ECOG >/-2)
5. Total bilirubin >1.8, creatinine >2, hemoglobin <10, platelets <50,000, WBC <2,000)
6. Active interstitial lung disease; asthma requiring more than as needed bronchodilators for management; or other autoimmune lung disease
7. Pregnancy (urine hCG)
8. Breast feeding
9. History of autoimmune disease
10. Involved in other experimental protocols (except with permission of the other study PI)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female or male
* Menopausal status not specified
* Immunologically intact by recall anergy testing
* Negative pregnancy test

Exclusion criteria:

* Karnofsky 0-60% or ECOG ≥ 2
* Total bilirubin > 1.8 g/dL
* Creatinine > 2.0 g/dL
* Hemoglobin < 10.0 g/dL
* Platelet count < 50,000/mm³
* WBC< 2,000/mm³
* Active pulmonary disease requiring medication that includes multiple inhalers
* Pregnancy
* Breastfeeding
* History of autoimmune disease

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics

Exclusion criteria:

* Concurrent immunosuppressive therapy including chemotherapy, steroids, or methotrexate
* Concurrent participation in another experimental treatment (except with permission of the other study investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2007-01; Primary Completion 2014-12-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Disease recurrence | Five years (from date of enrollment to the study through the end of the follow-up period)
  The following will be compared:
  1. disease recurrence rates between HLA-A2-negative patients receiving the AE37 + GM-CSF vaccine and HLA-A2-negative patients receiving GM-CSF alone
  2. disease recurrence rates between HLA-A2-positive patients receiving the GP2 + GM-CSF vaccine and HLA-A2-positive patients receiving GM-CSF alone
  3. disease recurrence rates between all four arms of the trial.

SECONDARY OUTCOMES:
Safety | Local and systemic reactions to each inoculation will be monitored every six months during the regular inoculation series and the booster series.
  Inoculations will be immediately halted if any serious adverse reactions occur which, when based upon appropriate judgment of the PI, are determined to jeopardize the patient or require medical or surgical intervention. Any death or grade 4 adverse drug experience found to be directly related to the experimental vaccine will result in suspension of patient enrollment to the study.
Immune Response | Immune response will be measured after every monthly inoculation in the regular inoculation series and after each inoculation in the booster series
  Immune response will be measured by proliferation assays, dimer assays, and ELISPOT. Delayed type hypersensitivity reactions will be compared between the vaccinated group and GM-CSF-only group.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Mittendorf, MD, FACS, Principal Investigator — UT M.D. Anderson Cancer Center; George E Peoples, MD, FACS, Study Director — Cancer Vaccine Development Program, Department of Surgery, Brooke Army Medical Center
Locations (13):
- United States (11):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Good Samaritan Hospital Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - San Antonio Army Medical Center, Fort Sam Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - STOH Clinical Research, San Antonio, Texas
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
- Landstuhl Regional Medical Center, Landstuhl, Kirchberg, Germany
- Saint Savas Cancer Hospital of Athens, Athens, Greece

REFERENCES:
- [Background] Mittendorf EA, Alatrash G, Xiao H, Clifton GT, Murray JL, Peoples GE. Breast cancer vaccines: ongoing National Cancer Institute-registered clinical trials. Expert Rev Vaccines. 2011 Jun;10(6):755-74. doi: 10.1586/erv.11.59. PMID 21692698
- [Result] Sears AK, Perez SA, Clifton GT, Benavides LC, Gates JD, Clive KS, Holmes JP, Shumway NM, Van Echo DC, Carmichael MG, Ponniah S, Baxevanis CN, Mittendorf EA, Papamichail M, Peoples GE. AE37: a novel T-cell-eliciting vaccine for breast cancer. Expert Opin Biol Ther. 2011 Nov;11(11):1543-50. doi: 10.1517/14712598.2011.616889. Epub 2011 Sep 6. PMID 21895539
- [Derived] Jackson DO, Trappey FA, Clifton GT, Vreeland TJ, Peace KM, Hale DF, Litton JK, Murray JL, Perez SA, Papamichail M, Mittendorf EA, Peoples GE. Effects of HLA status and HER2 status on outcomes in breast cancer patients at risk for recurrence - Implications for vaccine trial design. Clin Immunol. 2018 Oct;195:28-35. doi: 10.1016/j.clim.2018.06.008. Epub 2018 Jul 17. PMID 30025819
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://web.archive.org/web/20111026180718/http://cancer.gov/clinicaltrials/search/view?cdrid=562261&version=healthprofessional